CLINICAL TRIAL: NCT03504839
Title: Same Day Subcutaneous ICD And Send Home
Brief Title: Same Day Subcutaneous ICD And Send Home (DASH)
Acronym: DASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emile Daoud, MD (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Emile Daoud, MD, Sub-Investigator, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017H00451
Record Dates: First submitted 2018-04-04; First posted 2018-04-20 (Actual); Results first posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Cardiomyopathies; Cardiac Death, Sudden
Keywords: defibrillator
MeSH Terms: conditions — Cardiomyopathies; Death, Sudden, Cardiac

STUDY DESIGN:
Intervention Model Description: Consecutive patients consented for SICD as per standard indications for device implantation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention (Other): S-ICD implantation.
  Interventions: Device: Subcutaneous ICD with same day discharge

INTERVENTIONS:
Device: Subcutaneous ICD with same day discharge — Receiving a SICD and discharged the same day

SUMMARY:
Design: Prospective, non-randomized single center study at The Ohio State University Wexner Medical Center.

Purpose: The purpose of this study is to prospectively evaluate a specific analgesia protocol designed to allow for same day discharge following implantation of the subcutaneous implantable cardiac defibrillator (S-ICD) Enrollment: Up to 40 subjects will be enrolled. Subject Population: Consecutive patients undergoing S-ICD implantation under general anesthesia or monitored anesthesia care.

Endpoints: Rate of successful completion of the protocol; Procedural complications; Serial assessment of patient perception of pain.

DETAILED DESCRIPTION:
This is a prospective, nonrandomized, descriptive, single center study designed to assess the rate of successful completion of the study protocol in consecutive patients undergoing S-ICD implantation.

Objectives To prospectively evaluate the same day discharge protocol for patients undergoing S-ICD implantation.

Primary Endpoint 1. Rate of successful completion of S-ICD implantation and discharge of the patient on the same day the device is implanted using the analgesia protocol.

Secondary Endpoints

1. Procedure complication (failed implantation, infection, hematoma/bleeding, etc…) within 30 days of procedure.
2. Serial assessment of patient perception of pain using the graded integer pain scale of 1-10
3. Side effects related to medical therapy of protocol.
4. Time from beginning of recovery (defined as when the patient enters the recovery IPR room) to the time of discharge from the recovery unit.
5. 30 day readmission rate after discharge following S-ICD implant
6. Number of days that oral analgesics are used post discharge.

Patients will be approached for participation in the study once they have been consented for implantation of the clinically indicated S-ICD

.

Pre-procedure analgesia will be given to each patient as follows:

Acetaminophen 975 mg PO x 1 will be administered 1-2 hours prior to the procedure. and Oxycodone 10 mg PO x 1 will be administered 1-2 hours prior to the procedure. Anesthesia will be provided by anesthesiology team as MAC or general anesthesia. Local subcutaneous anesthetic will be a 50:50 mixture of 2% lidocaine and 0.5% bupivacaine; which will result in a concentration of 1% lidocaine and 0.25% bupivacaine.

Starting at ≈2 hours post procedure, the patient will then enter the "Preparation for Discharge" phase. The modified Aldrete scoring system will be used to determine eligibility for discharge home.Patients with an Aldrete score ≥ 9 will be deemed eligible for discharge home.

Additional standard ambulatory discharge criteria per the OSUWMC postanesthesia care policy statement will be applied by the nursing team, akin to all ambulatory surgery patients at OSUWMC. If the above discharge parameters (DP) are not meet, the patient will be reassessed every 30 minutes until parameters are satisfied. Once the patient satisfies the DP, the patient will complete the Pain Perception Questionnaire and be assessed for ambulation, eating/drinking and for understanding of post discharge instructions. The electrophysiology device nursing staff will review management of the S-ICD incision, device and post discharge care instructions with the patient and with the accompanying family member(s)/friend. The patient will be given instructions regarding management of pain and will be provided the following prescription for outpatient pain control Percocet 5mg/325 mg (1 tablet every 6 hours). A 2-day supply will be given.

Also, the patient will be provided a phone number to contact during business hours as well as for after hours to address questions/concerns.

The electrophysiology nursing staff will contact the patient the following day and again at about 3 days post discharge to administer the Pain Perception Questionnaire as well as to address any patient questions. The patient will then be evaluated in the Device Clinic about 10 days post implantation. The Pain Perception questionnaire will be administered and assessment of the incision and S-ICD will be completed. The last Pain Perception questionnaire will be obtained by telephone at about 30 days post implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient consented for implantation of S-ICD.
* Ambulatory/outpatient patient coming to the hospital setting solely for implantation of S-ICD
* Patient agrees to participate and is able to comply with the defined study protocol, including assistance for home care and transportation for the first ≈12-18 hours post discharge, and compliance with the required follow up.

Exclusion Criteria:

* Inability or unwillingness to provide informed consent
* Patients who, for any reason, was hospitalized or in an emergency department the day prior to the S-ICD implantation, including patients transferred for S-ICD implantation
* Patients in which the hemodynamics are dependent upon intravenous pressors infusing at the time of device implantation or mechanical support, inclusive of left ventricular assist device and intravenous devices (balloon pump, Impella device).
* Age < 18 years.
* Pregnancy.
* Currently incarcerated.
* Hypoxia (room air oxygen <91%) or acutely short of breath.
* Hypotension (Systolic blood pressure <90) unless this is patient's typical blood pressure).
* Bradycardia (heart rate <45bpm, unless this is patient's typical resting heart rate).
* Acute electrolyte disorder that cannot be easily corrected (e.g., potassium supplementations) based upon Chem 6 values obtained on day of procedure.
* Presence of a fever.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toshimasa Okabe, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 53
Completed | 49
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Rate of Successful Completion of S-ICD Implantation and Discharge of the Patient on the Same Day the Device is Implanted Using the Analgesia Protocol.
Description: Rate of successful completion of S-ICD implantation and discharge of the patient on the same day the device is implanted using the analgesia protocol.
Time Frame: within 30 days of the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 53
Participants | 49

2. Secondary Outcome: Procedure Complication (Failed Implantation, Infection, Hematoma/Bleeding, Etc…) Within 30 Days of Procedure.
Description: Procedure complication (failed implantation, infection, hematoma/bleeding, etc…) within 30 days of procedure.
Time Frame: within 30 days of the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 53
Participants | 4
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority; p < 0.01, ANOVA

3. Secondary Outcome: Serial Assessment of Patient Perception of Pain Using the Graded Integer Pain Scale of 0-10
Description: Serial assessment of patient perception of pain using the graded integer Numeric Pain Rating Scale (NPRS) of 0-10. This is an unidimensional measure of pain intensity in adults. Zero being no pain, 1-3 being mild pain, 4-6 being moderate pain, 7-10 being severe pain.
Time Frame: within 30 days of the procedure
Population: Patient's did not always answer/call back for their follow-up phone calls.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 49
Participants
  Post-Operation Day #0: mild pain | 37
  Post-Operation Day #0: moderate pain | 5
  Post-Operation Day #0: severe pain | 7
  Post-Operation Day #1: mild pain | 31
  Post-Operation Day #1: moderate pain | 11
  Post-Operation Day #1: severe pain | 7
  Post-Operation Day #3: number analyzed (Participants) | 48
  Post-Operation Day #3: mild pain | 39
  Post-Operation Day #3: moderate pain | 5
  Post-Operation Day #3: severe pain | 4
  Post-Operation Day #14: number analyzed (Participants) | 47
  Post-Operation Day #14: mild pain | 44
  Post-Operation Day #14: moderate pain | 1
  Post-Operation Day #14: severe pain | 2
  Post-Operation Day #30: number analyzed (Participants) | 48
  Post-Operation Day #30: mild pain | 46
  Post-Operation Day #30: moderate pain | 1
  Post-Operation Day #30: severe pain | 1

4. Secondary Outcome: Side Effects Related to Medical Therapy of Protocol.
Description: Side effects related to medical therapy of protocol.
Time Frame: within 30 days of the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 49
Participants | 0

5. Secondary Outcome: Time From Beginning of Recovery (Defined as When the Patient Enters the Recovery IPR Room) to the Time of Discharge From the Recovery Unit.
Description: Time from beginning of recovery (defined as when the patient enters the recovery IPR room) to the time of discharge from the recovery unit.
Time Frame: within 30 days of the procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intervention
Number analyzed (Participants) | 49
minutes | 534 (80)

6. Secondary Outcome: 30 Day Readmission Rate After Discharge Following S-ICD Implant
Description: 30 day readmission rate after discharge following S-ICD implant
Time Frame: within 30 days of the procedure
Population: There were 2 unplanned healthcare visits within 30 days of implantation conclusively related to S-ICD implantation due to incisional infection successfully treated with oral antibiotics and inappropriate shocks due to oversensing, leading to S-ICD removal. Neither of these complications, however, would have been prevented even if they had stayed overnight in the hospital following outpatient S-ICD implantation.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 49
Participants | 2

7. Secondary Outcome: Number of Days That Oral Analgesics Are Used Post Discharge.
Description: Number of days that oral analgesics are used post discharge.
Time Frame: within 30 days of the procedure
Measure: Number; unit: days
Arm/Group | Intervention
Number analyzed (Participants) | 49
days | 3

ADVERSE EVENTS:
Time Frame: 1 year, 3 months.
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 2/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=49)
Incisional infection (Infections and infestations) | 1 (1) — Incisional infection successfully treated with oral antibiotics.
Inappropriate S-ICD shocks (Cardiac disorders) | 1 (1) — Inappropriate shocks due to oversensing, leading to S-ICD removal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/39/NCT03504839/Prot_SAP_003.pdf
  • Informed Consent Form (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT03504839/ICF_000.pdf